CLINICAL TRIAL: NCT04734171
Title: COVID-19 and Its Implications on Social Activity, Loneliness and Stigma
Brief Title: Social Activity, Loneliness and Stigma During COVID-19 Outbreak
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Linda Valeri, Assistant Professor of Biostatistics, Department of Biostatistics, Columbia University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: AAAT0067
Record Dates: First submitted 2021-01-29; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Covid19; Fear; Loneliness
Keywords: Covid19 related stigma, fear and loneliness
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Informational sheet (IS) (Placebo Comparator): participant receives an informational sheet about COVID-19
  Interventions: Behavioral: Informational sheet
- IS + Video Solo (Active Comparator): participants an informational sheet about COVID-19 and a 90 seconds video aimed at sensitizing participants to COVID-19 related stigma
  Interventions: Behavioral: Informational sheet; Behavioral: Stigma awareness video intervention
- IS + Video Friends (Active Comparator): participants an informational sheet about COVID-19 and a 150 seconds video aimed at encouraging the use of a digital device (i.e. not in person contact) to meet with friends.
  Interventions: Behavioral: Digital social activity video intervention; Behavioral: Informational sheet
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Digital social activity video intervention — A 150 seconds video aimed at encouraging the use of a digital device (i.e. not in person contact) to meet with friends during the COVID-19 pandemic. Two friends meet via zoom instead of in person and share their experiencing supporting each other.
  Arms: IS + Video Friends
Behavioral: Informational sheet — An informational sheet to learn about the COVID-19 outbreak (standard).
  Other Names: Vignette
  Arms: IS + Video Friends; IS + Video Solo; Informational sheet (IS)
Behavioral: Stigma awareness video intervention — A video aimed at sensitizing participants to COVID-19 related stigma. A COVID-19 + individual share their experience.
  Arms: IS + Video Solo

SUMMARY:
The overall goal of this study is to evaluate the association of quarantine measures for COVID-19 and perceived anxiety, stigma and loneliness and to evaluate the efficacy of interventions in reducing anxiety, loneliness and perception of stigma induced by self-isolation during the outbreak.

Specific Aims:

In the proposed study, participants will include members of the United States general population who will be randomly assigned to either (a) a vignette to learn about the COVID-19 outbreak, (b) a vignette to learn about the COVID-19 outbreak AND a video aimed at encouraging the use of a digital device (i.e. not in person contact) to meet with friends, (c) a vignette to learn about the COVID-19 outbreak AND a video aimed at sensitizing participants to COVID-19 related stigma, (d) Control arm. Web-based self-report questionnaires will be conducted to compare interventions and control groups. The short and low-cost online module will allow recruitment of a large sample of people.

Hypotheses:

(1) the video-based intervention groups will demonstrate lower rates of anxiety and loneliness than vignette and control groups, (2) the video-based group that presents an individual with COVID-19 will demonstrate lower rate of stigma than other groups.

DETAILED DESCRIPTION:
Currently, the world is experiencing a Coronavirus outbreak, COVID-19, which originated in mainland China in December 2019, spread rapidly to South Korea and Europe, Italy in particular, between January and March of 2020 and is currently spreading in all continents and has been recognized as a pandemic. It is of high importance to monitor how the trends in COVID-19 outbreak are shaping the social contexts and norms across communities and families. In a time in which individuals all over the world are experiencing quarantine, it is important to evaluate the potential surge of the phenomena of social anxiety, stigma, and of perceived fear and loneliness. Furthermore, it is critical to study interventions that aim to reduce each of these. The overall goal of this study is to evaluate the association of quarantine measures for COVID-19 and perceived anxiety, stigma and loneliness and to evaluate the efficacy of interventions in reducing anxiety, loneliness and perception of stigma induced by self-isolation during the outbreak. The hypotheses will be tested using ANOVA and multinomial logistic regressions. An alpha level of 0.01 will be used to account for multiple testing.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Younger than 70 years old
* United States resident

Exclusion Criteria:

* Less than 18 years old

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2020-04-16 (Actual); Study Completion 2020-04-16 (Actual)

PRIMARY OUTCOMES:
Change in total stigma score 2 weeks after the intervention | Baseline and 2 weeks
  This is designed to measure stigma associated with COVID-19. A continuous variable will be obtained as a sum of questionnaire items ordinal answers (4 questions, score range 4-16, 4 = low stigma, 16 = high stigma) adapted from the HIV stigma validated questionnaire (HIV stigma scale, Berger et al., 2001).
  1. Strongly disagree = 1
  2. Disagree = 2
  3. Agree = 3
  4. Strongly agree = 4
  5. prefer not to answer: missing value
Change in total fear score 2 weeks after the intervention | Baseline and 2 weeks
  This is designed to measure fear associated with COVID-19. A continuous variable will be obtained as a sum of questionnaire items (4 questions, score range 4-16, 4 = low fear, 16 = high fear) addressing fear of contracting COVID-19 and fear of consequences of COVID-19.
  1. Not at all = 1
  2. A bit = 2
  3. Quite a bit = 3
  4. A lot = 4
  OR
  1. Strongly disagree = 1
  2. Disagree = 2
  3. Agree = 3
  4. Strongly agree = 4
  5. Prefer not to answer = missing value
Change in loneliness ordinal score 2 weeks after the intervention | Baseline and 2 weeks
  Subjects will answer the following questionnaire item and an ordinal variable will be calculated (1 = low loneliness, 4 = high loneliness):
  How lonely do you feel?
  1. Not at all = 1
  2. A bit = 2
  3. Quite a bit = 3
  4. A lot = 4
Change in fear of people COVID-19+ ordinal score 2 weeks after the intervention | Baseline and 2 weeks
  Ordinal variable from the questionnaire item (1 = low fear of people, 4 = high fear of people):
  How much are you afraid of people diagnosed with Coronavirus (COVID-19)?
  1. Not at all = 1
  2. A bit = 2
  3. Quite a bit = 3
  4. A lot = 4

SECONDARY OUTCOMES:
Change in time spent on internet ordinal score 2 weeks after the intervention | Baseline and 2 weeks
  Ordinal variable from the questionnaire item time spent on the internet (for leisure or work-related activities) in the past week (averaged in number of hours)(1 = less time, 4 = more time):
  1. <1 h = 1
  2. 1h-4h = 2
  3. 4h-7h = 3
  4. >7h = 4
Change in social activity ordinal score 2 weeks after the intervention | Baseline and 2 weeks
  Ordinal variable from the questionnaire item on social contact seeking behavior in the past week (How many times did you contact [in person or via video call] your friends/family members over the last week (1 = low social activity, 4 = high social activity)?
  1. 0-2 = 1
  2. 2-5 = 2
  3. 5-7 = 3
  4. more than 7 = 4

CONTACTS AND LOCATIONS:
Overall Officials: Linda Valeri, PhD, Principal Investigator — Assistant Professor of Biostatistics
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No